CLINICAL TRIAL: NCT00003211
Title: Treatment of Newly Diagnosed Medulloblastoma and Supratentorial PNET in Patients At Least 3 Years With a Phase II Topotecan Window (High-Risk Patients Only), Risk-Adapted Radiation Therapy, and Dose-Intensive Chemotherapy With Peripheral Blood Stem Cell Support
Brief Title: Chemotherapy, Radiation Therapy, and Peripheral Stem Cell Transplantation in Treating Children With Newly Diagnosed Medulloblastoma or Supratentorial Primitive Neuroectodermal Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000066069; SJCRH-MB-96 (Other: St. Jude Children's Research Hospital); SJMB-96 (Other: St. Jude Children's Research Hospital); NCI-G98-1387 (Other: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2003-07-09 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-11

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Filgrastim; Amifostine; Cisplatin; Cyclophosphamide; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Average-risk (Experimental): Participants meeting the eligibility requirements for assignment to the average-risk arm.
  Interventions: filgrastim, amifostine trihydrate, cisplatin, cyclophosphamide, vincristine sulfate, peripheral blood stem cell transplantation, radiation therapy.
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: cisplatin; Drug: cyclophosphamide; Drug: vincristine sulfate; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy
- High-risk (Experimental): Participants meeting the eligibility requirements for assignment to the high-risk arm.
  Interventions: filgrastim, amifostine trihydrate, cisplatin, cyclophosphamide, vincristine sulfate, peripheral blood stem cell transplantation, radiation therapy.
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: cisplatin; Drug: cyclophosphamide; Drug: vincristine sulfate; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
Drug: cisplatin
Drug: cyclophosphamide
Drug: vincristine sulfate
Procedure: peripheral blood stem cell transplantation
  Other Names: PBSCT
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy and radiation therapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy or radiation therapy and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy with topotecan, cyclophosphamide, cisplatin, and vincristine plus radiation therapy and peripheral stem cell transplantation in treating children with newly diagnosed medulloblastoma or supratentorial primitive neuroectodermal tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Estimate the response rate to topotecan in children with newly diagnosed medulloblastoma or supratentorial primitive neuroectodermal tumors who have measurable residual disease after surgery. (Topotecan window closed to accrual 9/10/2001)
* Determine the feasibility of four courses of high-dose chemotherapy (vincristine, cisplatin, and cyclophosphamide) with peripheral blood stem cell support after craniospinal irradiation (CSI) in these patients.
* Estimate the 5-year overall survival and progression-free survival in patients treated with risk-adapted CSI and high-dose chemotherapy.
* Compare changes in intellectual functioning in patients treated with reduced-dose vs standard-dose CSI.
* Estimate the incidence of ototoxicity associated with risk-adapted CSI and posterior fossa boost(s) given by 3-D conformal radiotherapy technique combined with amifostine and cisplatin.

OUTLINE: This is a multicenter study. Patients are assigned to 1 of 2 treatment groups based on risk status.

* Group 1 (average-risk): Patients receive filgrastim (G-CSF) subcutaneously (SC) or IV daily until peripheral blood stem cells (PBSC) are harvested. PBSC are harvested when blood counts recover. Patients then receive craniospinal irradiation (CSI) 5 days a week for 6 weeks. Beginning 6 weeks after completion of CSI, patients receive high-dose chemotherapy comprising vincristine IV followed by cisplatin IV over 6 hours on day -4 and cyclophosphamide IV over 1 hour on days -3 and -2. Patients receive amifostine IV over 1 minute a maximum of 5 minutes prior to cisplatin infusion and then 3 hours into cisplatin infusion. PBSC are reinfused on day 0. Patients receive G-CSF SC beginning on day 1 and continuing for a minimum of 7 days or until blood counts recover. Vincristine IV is administered on day 6. G-CSF is stopped 48 hours prior to beginning subsequent courses of chemotherapy. High-dose chemotherapy repeats every 4 weeks for 4 courses.
* Group 2 (high-risk): Patients receive topotecan IV over 4 hours on days 1-5 and G-CSF SC or IV beginning 24 hours after completion of the first course of topotecan and continuing until PBSC are harvested. Treatment repeats every 3 weeks for 2 courses. If an adequate number of PBSC are not harvested, the patient undergoes a second harvest of PBSC after the second course of topotecan. Patients then receive CSI, high-dose chemotherapy, amifostine, and PBSC support as in group 1. (Topotecan window closed to accrual 9/10/2001) Patients undergo neuropsychological testing prior to radiotherapy and chemotherapy and then at 1, 2, and 5 years.

Patients are followed at 1, 2, 4, 6, 9, 12, 15, 18, and 24 months and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 12-36 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven medulloblastoma or supratentorial primitive neuroectodermal tumor
* Average-risk group:

  * Localized tumor with no overt evidence of invasion beyond the posterior fossa
  * Less than 1.5 cm2 residual tumor/imaging abnormality
  * No CNS or extraneural metastasis (confirmed by bone scan)
  * Brain stem invasion allowed if above criteria met
* High-risk group:

  * Metastatic disease within the neuraxis (subarachnoid dissemination) OR greater than 1.5 cm^2 residual disease at the primary site after surgery
* No bone involvement by bone scan
* Must begin study within 28 days of definitive surgery

PATIENT CHARACTERISTICS:

Age

* 3 to 20 at diagnosis

Performance status

* ECOG 0-3 (except patients with posterior fossa syndrome)

Life expectancy

* Not specified

Hematopoietic

* WBC greater than 3,000/mm^3
* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 10 g/dL

Hepatic

* Bilirubin less than 1.5 mg/dL
* SGPT less than 1.5 times normal

Renal

* Creatinine less than 1.2 mg/dL OR
* Creatinine clearance greater than 70 mL/min

Other

* Not pregnant or nursing
* Negative pregnancy test
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Prior corticosteroids allowed

Radiotherapy

* No prior radiotherapy

Surgery

* See Disease Characteristics

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 94 (Actual)
Dates: Start 1996-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, MD, Study Chair — St. Jude Children's Research Hospital
Locations (4):
- United States (2):
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center, Houston, Texas
- Australia (2):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Parkville, Victoria

REFERENCES:
- [Result] Laughton SJ, Merchant TE, Sklar CA, Kun LE, Fouladi M, Broniscer A, Morris EB, Sanders RP, Krasin MJ, Shelso J, Xiong Z, Wallace D, Gajjar A. Endocrine outcomes for children with embryonal brain tumors after risk-adapted craniospinal and conformal primary-site irradiation and high-dose chemotherapy with stem-cell rescue on the SJMB-96 trial. J Clin Oncol. 2008 Mar 1;26(7):1112-8. doi: 10.1200/JCO.2008.13.5293. PMID 18309946
- [Result] Gajjar A, Chintagumpala M, Ashley D, Kellie S, Kun LE, Merchant TE, Woo S, Wheeler G, Ahern V, Krasin MJ, Fouladi M, Broniscer A, Krance R, Hale GA, Stewart CF, Dauser R, Sanford RA, Fuller C, Lau C, Boyett JM, Wallace D, Gilbertson RJ. Risk-adapted craniospinal radiotherapy followed by high-dose chemotherapy and stem-cell rescue in children with newly diagnosed medulloblastoma (St Jude Medulloblastoma-96): long-term results from a prospective, multicentre trial. Lancet Oncol. 2006 Oct;7(10):813-20. doi: 10.1016/S1470-2045(06)70867-1. PMID 17012043
- See also: St. Jude Children's Research Hospital — http://www.stjude.org